CLINICAL TRIAL: NCT00154648
Title: An Open, Contrast-Enhanced Magnetic Resonance Angiography (CE-MRA) Study of Arteries Using Gadovist 1.0 in Comparison to Intra-Arterial Digital Subtraction Angiography (IA DSA) Using Ultravist
Brief Title: CE-MRA Using Gadovist in Comparison to IA DSA Using Ultravist
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0941540200
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2005-06

CONDITIONS: Angiography, Digital Subtraction; Magnetic Resonance Angiography
Keywords: MRA; DSA; gadovist; angiography

INTERVENTIONS:
Procedure: CE-MRA

SUMMARY:
This trial is to show the diagnostic efficacy of Gadovist for contrast enhanced magnetic resonance angiography (CE-MRA) of the arteries.

DETAILED DESCRIPTION:
This trial is to show the diagnostic efficacy of Gadovist for contrast enhanced Magnetic Resonance Angiography (CE-MRA) of arteries (specified vessel segments) by analyzing the rate of agreement, image quality, and diagnostic confidence between a CE-MRA based diagnosis and the diagnosis achieved from the comparator procedure IA DSA using Ultravist.

ELIGIBILITY:
Inclusion Criteria:

* With suspected or known disease of the arteries
* Scheduled for an IA DSA/cut film angiography of the arteries in a period of less than 7 days prior to or after the study period and has completed delineation and documentation of all vessels.
* Willing and able to continue study participation. This includes the administration of Gadovist® 1.0 and completion of all procedures required by the study protocol
* Patient is between 20 and 75 years of age
* Fully informed and has signed consent in advance

Exclusion Criteria:

* Patient is clinically unstable or his/her clinical course during the 72 hour safety observation period was unpredictable
* Patient with renal failure
* Woman who is pregnant or of childbearing potential without having had a negative pregnancy test prior to enrollment (within 72 hours prior to CE-MRA)
* Lactating woman
* Patient with any contraindication to magnetic resonance imaging (MRI) examination and IA DSA.
* Patient receives any investigational drug within 30 days prior to study entry or is planned to receive any other investigational drug during the safety follow-up (72 hours after CE-MRA).
* Patient is scheduled for surgery or other interventions within the 72 hours after the CE-MRA/IA DSA or had any such procedure within 48 hours prior to the study CE-MRA/IA DSA.
* Hypersensitivity to gadobutrol products
* Patient has previously entered this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-06

PRIMARY OUTCOMES:
Rate of agreement
Image quality
Diagnostic confidence

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Man Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan